CLINICAL TRIAL: NCT06169293
Title: Evaluation of an Interactive Mental Wellness (I-AM-WELL) Program on Final Year Nursing Students: A Mixed Methods Evaluation
Brief Title: Evaluation of an Interactive Mental Wellness (I-AM-WELL) Program on Final Year Nursing Students
Acronym: I-AM-WELL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NUS-IRB-2023-641
Record Dates: First submitted 2023-12-01; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Resilience; Practice Readiness; Depression; Anxiety; Stress; Physical Activity; Eating Behavior
MeSH Terms: conditions — Depression; Anxiety Disorders; Motor Activity; Feeding Behavior

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-AM-WELL program (Experimental)
  Interventions: Behavioral: I-AM-WELL
- Waitlist control (No Intervention): Students will receive the intervention after data is collected from all three time points

INTERVENTIONS:
Behavioral: I-AM-WELL — The I-AM-WELL program adopts an asynchronous online learning approach and will be delivered over one week by a trained counsellor, and a nurse researcher.
  Students will attend an online self-paced program. The program will comprise of topics such as: (1) Resilience and protective factors, (2) introduction to clinical nursing education, (3) experiences of clinical attachments, and (4) stress, physical wellbeing and diet materials. Students will have access to online materials (e.g., short videos), have opportunities to discuss (e.g., forum) and infographics.
  Overall, the program will be delivered over in one week lasting six hours.
  Arms: I-AM-WELL program

SUMMARY:
This study aims to address the following research questions:

Evaluate the effectiveness of an Interactive Mental Wellness (I-AM-WELL) program on final year nursing students' anxiety, depression, stress, resilience, practice readiness, physical activity and eating behaviours.

Explore final year nursing students' experiences and perception of the I-AM-WELL program.

Participants will be invited to participate in an asynchronous online I-AM-WELL program

ELIGIBILITY:
Inclusion Criteria:

* Final year nursing students enrolled in the undergraduate nursing program
* Above the ages of 18 years
* Able to comprehend the English language
* Have a device that can connect to the Internet

Exclusion Criteria:

* Students who refused to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-25 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Resilience | Before training
  Brief Resilience Scale
Resilience | Immediately after training
  Brief Resilience Scale
Depression, Anxiety and Stress | Before training
  Depression, Anxiety and Stress Scale - 21
Depression, Anxiety and Stress | Immediately after training
  Depression, Anxiety and Stress Scale - 21
Practice Readiness | Before training
  Nursing Practice Readiness Scale
Practice Readiness | Immediately after training
  Nursing Practice Readiness Scale
Physical Activity | Before training
  International Physical Activity Questionnaire
Physical Activity | Immediately after training
  International Physical Activity Questionnaire
Eating behaviours | Before training
  Self-regulation of eating behaviours scale
Eating behaviours | Immediately after training
  Self-regulation of eating behaviours scale

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Ang, PhD, Principal Investigator — National University of Singapore

IPD SHARING:
Plan to Share IPD: Undecided